CLINICAL TRIAL: NCT06571890
Title: Emergence Agitation in Paediatric Day Care Surgery: A Randomised, Single-blinded Study Comparing Narcotrend and Heart Rate Variability With Standard Monitoring
Brief Title: Emergence Agitation in Paediatric Day Care Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense Patient Data Explorative Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 280482
Record Dates: First submitted 2024-04-02; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Delirium; Postoperative Agitation; Anesthesia; Pain Monitoring; Heart Rate Variability; Narcotrend; Mdoloris; Anesthesia Nociception Index
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard (STD) (No Intervention): Standard anaesthesia with Sevoflurane Inhalation anaesthesia, fentanyl and a laryngeal mask
- Narcotrend (NCT) (Experimental): Standard anaesthesia with Sevoflurane inhalation anaesthesia, fentanyl and a laryngeal mask. Sevoflurane concentration was titrated via a Narcotrend bispectral anaesthesia monitor.
  Interventions: Device: Narcotrend bispectral index anaesthesia monitor
- Anaesthesia Nociception Index Monitor (ANI) (Experimental): Standard anaesthesia with Sevoflurane inhalation anaesthesia, fentanyl and a laryngeal mask. Fentanyl dosage titrated with guidance from Mdoloris ANI monitor, a heart rate variability-based nociception monitor. When a threshold value is exceeded, additional fentanyl 1 mcg/kg is given
  Interventions: Device: Mdoloris Anaesthesia Nociception Monitor

INTERVENTIONS:
Device: Narcotrend bispectral index anaesthesia monitor — A bispectral index anaesthesia monitor collects simplified EEG via forehead electrodes and displays an index of 0-100, where an index of 40-60 is considered optimal
  Arms: Narcotrend (NCT)
Device: Mdoloris Anaesthesia Nociception Monitor — A heart rate variability-based nociception monitor collects ECG-signal from electrodes on the patient's chest and displays an index of 0-100 where an index below 50 is considered nociceptive.
  Arms: Anaesthesia Nociception Index Monitor (ANI)

SUMMARY:
Emergence agitation is a significant and persistent challenge in paediatric anaesthesia, especially in children of preschool age.

In this study, the investigators examined whether anaesthesia titration with either a sleep depth monitor or a pain monitor would result in changed postoperative agitation rates, measured via the Richmond Agitation and Sedation Score (RASS).

93 children participated. The participants were divided into three groups: A conventional anaesthesia group, an EEG (Electroencephalography)- monitored and a pain-monitored group. The pain-monitored children received the most pain medication but were discharged at the same rate as the other children with unchanged rates of nausea and vomiting and less agitation than the sleep-monitored children.

DETAILED DESCRIPTION:
Healthy preschool outpatients assigned for abdominal/inguinal hernia and cryptorchidism repairs participated after parental consent.

One group received standard anaesthesia induction and maintenance, according to the usual ward regimen. This was done with sevoflurane inhalation, fentanyl bolus and a laryngeal mask airway (Standard group, STD group)

The second group received standard anaesthesia as well only this time the sevoflurane titration was guided via the Nacotrend bispectral index monitor, towards a narcotrend index of 2-4. (Narcotrend group, NCT group)

The third group also received standard anaesthesia and was additionally monitored with a Mdoloris Anaesthesia Nociception Index (ANI) monitor for perioperative nociception. When a nociceptive threshold was exceeded, an extra bolus of fentanyl of 1 mcg/kg was given (ANI group)

All children were then escorted to the postoperative care unit for wakeup. A Richmond Agitation Sedation Scale score (RASS-score) was made every 15 minutes until discharge. This was analysed with Kaplan-Meyer mortality graph, along with usual statistics of secondary outcomes.

The children in the ANI group received the least fentanyl and were discharged no later than all the other children.

ELIGIBILITY:
Inclusion Criteria:

* Day surgery for abdominal and urological procedures
* Children 1-6 years
* American Society of Anesthesiologist (ASA) scale 1- 2
* Airway management with laryngeal masks or facemasks
* Consent from both parents/legal representatives
* Rescue propofol is allowed

Exclusion Criteria:

* Age less than 1 or older than 6 years
* ASA > 2
* Endotracheal intubation;
* Lack of consent from both parents/legal representatives
* Daily intake of medications that interfered with the autonomic nervous system reactivity, for example, inhaled beta-agonists for bronchial asthma and total intravenous anaesthesia (TIVA).

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Richmond Agitation Sedation Scale Score | During postoperative care unit (PACU) stay within 0-8 hours
  Scoring system for sedation and agitation from -5 til +4.

SECONDARY OUTCOMES:
Time consumption | Within 48 hours of hospital admission
  Time spent with anesthesia, PACU stay and total time.
Fentanyl consumption | Within 48 hours of hospital admission
  Given during the anesthesia against postoperative pain
Nurse-VAS | Within the duration of PACU stay of 0-8 hours
  A Visual-Analogue-Scale score (VAS score) assessed by PACU nurses. A score from 0-10 where 10 represents worst pain.
PONV | Within the duration of PACU stay of 0-8 hours
  Postoperative nausea and vomiting (PONV). A score from 0-2 where 2 represents worst nausea and vomiting.
Other medications | During the first 24 postoperative hours
  Other drugs, such as NSAIDs, given

CONTACTS AND LOCATIONS:
Overall Officials: Line Gry Larsen, Principal Investigator — Anaeshtesiologic Intensive Ward V, Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No